CLINICAL TRIAL: NCT01644396
Title: An Open-Label, Prospective Study to Assess the Safety and Effectiveness of Adalimumab (Humira®) in Patients With Moderate to Severe Plaque Psoriasis in the Russian Federation
Brief Title: An Open-Label, Prospective Study to Assess the Safety and Effectiveness of Adalimumab in Patients With Moderate to Severe Plaque Psoriasis in the Russian Federation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-279
Record Dates: First submitted 2012-05-07; First posted 2012-07-19 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Moderate to Severe Plaque Psoriasis
Keywords: Moderate to Severe Plaque Psoriasis
MeSH Terms: interventions — Adalimumab

ARMS (1):
- Adalimumab (Other): Participants received an initial adalimumab 80 mg subcutaneous dose, followed by adalimumab 40 mg subcutaneous every other week starting one week after the initial dose for up to 24 weeks.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab
  Other Names: ABT-D2E7; Humira

SUMMARY:
This is an open-label study designed to establish the safety and effectiveness of adalimumab in the treatment of moderate to severe plaque psoriasis after 24 weeks of treatment.

DETAILED DESCRIPTION:
During the treatment period, participants will receive an initial adalimumab 80 milligram (mg) subcutaneous (sc) dose, followed by adalimumab 40 mg sc every other week starting one week after initial dose. Safety and effectiveness assessments will be completed at Baseline, Week 2, Week 4, Week 8, Week 12, Week 16 and Week 24. Participants may discontinue adalimumab treatment at any time during study participation. Participants that end study participation early will have a Premature Discontinuation visit. All participants who do not initiate commercial Humira® will have a follow-up phone call 70 days after the last administration of study drug to obtain information on any new or ongoing Adverse Events (AEs). The 70-day follow-up phone call will not be required for any participant that initiates adalimumab therapy not supplied in the context of the clinical trial after the end of study participation.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for study participation if he/she meets the following criteria:

1. Male and female patients ≥ 18 years of age.
2. Clinical diagnosis of psoriasis for at least 6 months as determined by patient interview of his/her medical history and confirmation of diagnosis through physical examination by the investigator.
3. Stable plaque psoriasis for at least 2 months before Screening and Baseline visits as determined by patient interview of his/her medical history.
4. Moderate to severe plaque psoriasis defined by ≥ 10% Body Surface Area (BSA) involvement at the Baseline visit.
5. PASI (Psoriasis Area and Severity Index) score ≥ 10 at the Baseline visit.

Exclusion Criteria:

1. Diagnosis of erythrodermic psoriasis, pustular psoriasis, medication induced or medication-exacerbated psoriasis or new onset of guttate psoriasis.
2. Diagnosis of other active skin diseases or skin infections (bacterial, fungal, or viral) that may interfere with evaluation of psoriasis.
3. Patient who cannot discontinue topical therapies for the treatment of psoriasis such as corticosteroids, vitamin D analogs, or retinoids at least 14 days prior to the Baseline (Week 0) visit and during the study. Participants are allowed to use:

   * Shampoos that contain no corticosteroid;
   * Bland (without beta or alpha hydroxy acids or containing no psoriasis treatment) emollients;
   * Low potency topical corticosteroids on the palms, soles, face, inframammary area, and groin only.
4. Patient who cannot avoid UVB (Ultraviolet-B) phototherapy for at least 14 days prior to the Baseline (Week 0) visit and during the study.
5. Patient who cannot avoid PUVA (psoralen + ultraviolet A) phototherapy for at least 28 days prior to the Baseline (Week 0) visit and during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Okun, MD, Study Director — AbbVie
Locations (7):
- Russia (7):
  - Site Reference ID/Investigator# 78433, Kazan'
  - Site Reference ID/Investigator# 67542, Moscow
  - Site Reference ID/Investigator# 78413, Saint Petersburg
  - Site Reference ID/Investigator# 67545, Saint Petersburg
  - Site Reference ID/Investigator# 67546, Saratov
  - Site Reference ID/Investigator# 78417, Smolensk
  - Site Reference ID/Investigator# 67547, Yekaterinburg

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adalimumab
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population, defined as all enrolled participants who received at least 1 dose of adalimumab.
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 36
Region of Enrollment [Number; unit: participants]
  Russian Federation | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Psoriasis Area and Severity Index 75 (PASI 75) Response at Week 24
Description: The percentage of participants with a ≥ 75% reduction (improvement) in Psoriasis Area and Severity Index (PASI) score from Baseline. PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population; non-responder imputation (NRI) was used, where participants with a missing value were counted as a non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
percentage of participants | 82.0

2. Other Pre Specified Outcome: Change From Baseline in Hemoglobin
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: Intent-to-treat population; participants with non-missing Baseline and at least 1 post-baseline observation are included in the analysis.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
g/L | 0.6 (9.75)

3. Other Pre Specified Outcome: Change From Baseline in Hematocrit
Description: Safety variables included laboratory data, vital signs and adverse events. The hematocrit measures the volume of red blood cells compared to the total blood volume (red blood cells and plasma).
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters/liter
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
liters/liter | 0.007 (0.0348)

4. Other Pre Specified Outcome: Change From Baseline in Red Blood Cell Count
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: × 10^12 cells/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
× 10^12 cells/L | 0.02 (0.352)

5. Secondary Outcome: Percentage of Participants Achieving a Physician's Global Assessment of Clear
Description: The Physician's Global Assessment (PGA) is a 6-point scale used to measure the severity of disease at the time of the qualified investigator's evaluation of the participant. The degree of overall lesion severity was evaluated using the following categories:
  * 0: No evidence of scaling, erythema, or plaque elevation, overall score of cleared;
  * 1: Occasional fine scale over <5% of lesions, faint erythema, minimal plaque elevation, overall score of minimal;
  * 2: Fine scale dominates, light red coloration, mild plaque elevation, overall score of mild;
  * 3: Course scale dominates, moderate red coloration, moderate plaque elevation, overall score of moderate;
  * 4: Thick non-tenacious scale dominates, bright red coloration, marked plaque elevation, overall score of marked;
  * 5: Very thick tenacious scale predominates, dusky to deep red coloration, severe plaque elevation, overall score of severe.
  The percentage of participants achieving a PGA score of clear (0) is reported.
Time Frame: Weeks 2, 4, 8, 12, 16 and 24
Population: Intent-to-treat population; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
percentage of participants
  Week 2 | 0
  Week 4 | 0
  Week 8 | 6.0
  Week 12 | 20.0
  Week 16 | 60.0
  Week 24 | 70.0

6. Secondary Outcome: Percentage of Participants Achieving a Physician's Global Assessment of Clear or Minimal
Description: The Physician's Global Assessment (PGA) is a 6-point scale used to measure the severity of disease at the time of the qualified investigator's evaluation of the participant. The degree of overall lesion severity was evaluated using the following categories:
  * 0: No evidence of scaling, erythema, or plaque elevation, overall score of cleared;
  * 1: Occasional fine scale over <5% of lesions, faint erythema, minimal plaque elevation, overall score of minimal;
  * 2: Fine scale dominates, light red coloration, mild plaque elevation, overall score of mild;
  * 3: Course scale dominates, moderate red coloration, moderate plaque elevation, overall score of moderate;
  * 4: Thick non-tenacious scale dominates, bright red coloration, marked plaque elevation, overall score of marked;
  * 5: Very thick tenacious scale predominates, dusky to deep red coloration, severe plaque elevation, overall score of severe.
  The percentage of participants achieving a PGA score of clear (0) or minimal (1) is reported.
Time Frame: Weeks 2, 4, 8, 12, 16 and 24
Population: Intent-to-treat population; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
percentage of participants
  Week 2 | 2.0
  Week 4 | 12.0
  Week 8 | 34.0
  Week 12 | 72.0
  Week 16 | 86.0
  Week 24 | 80.0

7. Secondary Outcome: Percentage of Participants Achieving a One Grade Improvement in Physician's Global Assessment (PGA)
Description: The PGA is a 6-point scale used to measure the severity of disease at the time of the qualified investigator's evaluation of the participant. The degree of overall lesion severity was evaluated using the following categories:
  * 0: No evidence of scaling, erythema, or plaque elevation, overall score of cleared;
  * 1: Occasional fine scale over <5% of lesions, faint erythema, minimal plaque elevation, overall score of minimal;
  * 2: Fine scale dominates, light red coloration, mild plaque elevation, overall score of mild;
  * 3: Course scale dominates, moderate red coloration, moderate plaque elevation, overall score of moderate;
  * 4: Thick non-tenacious scale dominates, bright red coloration, marked plaque elevation, overall score of marked;
  * 5: Very thick tenacious scale predominates, dusky to deep red coloration, severe plaque elevation, overall score of severe.
  The percentage of participants achieving a shift from Baseline to a less severe category is reported.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16 and 24
Population: Intent-to-treat population; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
percentage of participants
  Week 2 | 40.0
  Week 4 | 74.0
  Week 8 | 98.0
  Week 12 | 98.0
  Week 16 | 100
  Week 24 | 96.0

8. Secondary Outcome: Percentage of Participants Achieving a PASI 50 Response
Description: The percentage of participants with a ≥ 50% reduction (improvement) in Psoriasis Area and Severity Index (PASI) score from Baseline. PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, and 24
Population: Intent-to-treat population; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
percentage of participants
  Week 2 | 8.0
  Week 4 | 36.0
  Week 8 | 84.0
  Week 12 | 88.0
  Week 16 | 94.0
  Week 24 | 96.0

9. Secondary Outcome: Percentage of Participants Achieving a PASI 75 Response
Description: as for outcome 1
Time Frame: Baseline and Weeks 2, 4, 8, 12, and 16
Population: Intent-to-treat population; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
percentage of participants
  Week 2 | 0
  Week 4 | 4.0
  Week 8 | 44.0
  Week 12 | 76.0
  Week 16 | 82.0

10. Secondary Outcome: Percentage of Participants Achieving a PASI 90 Response
Description: The percentage of participants with a ≥ 90% reduction (improvement) in Psoriasis Area and Severity Index (PASI) score from Baseline. PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, and 24
Population: Intent-to-treat population; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
percentage of participants
  Week 2 | 0
  Week 4 | 0
  Week 8 | 20.0
  Week 12 | 48.0
  Week 16 | 72.0
  Week 24 | 76.0

11. Secondary Outcome: Percentage of Participants Achieving a PASI 100 Response
Description: The percentage of participants with a 100% reduction (improvement) in Psoriasis Area and Severity Index (PASI) score from Baseline. PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, and 24
Population: Intent-to-treat population; non-responder analysis was used.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
percentage of participants
  Week 2 | 0
  Week 4 | 0
  Week 8 | 2.0
  Week 12 | 20.0
  Week 16 | 50.0
  Week 24 | 64.0

12. Secondary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Score
Description: PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
  Change from Baseline is presented as a percentage of the Baseline value: Post-baseline value - Baseline value / Baseline value * 100. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, and 24
Population: Intent-to-treat population; last observation carried forward (LOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
percent change
  Week 2 | -20.42 (15.586)
  Week 4 | -45.75 (17.444)
  Week 8 | -69.28 (20.759)
  Week 12 | -81.74 (25.039)
  Week 16 | -89.42 (19.789)
  Week 24 | -91.18 (16.579)

13. Secondary Outcome: Percent Change From Baseline in Dermatology Life Quality Index (DLQI)
Description: The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment related feelings. Participants answer 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is 0 to 30. A score of 21 to 30 means an extremely large effect on the participant's life whereas 0-1 means that the disease has no effect at all. Change from Baseline is presented as a percentage of the Baseline value: Post-baseline value - Baseline value / Baseline value * 100. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 8, 12, and 24
Population: Intent-to-treat population with available data; last observation carried forward (LOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 49
percent change
  Week 8 | -60.04 (40.435)
  Week 12 | -75.03 (45.311)
  Week 24 | -79.16 (34.784)

14. Secondary Outcome: Percent Change From Baseline in Nail Psoriasis Severity Index (NAPSI)
Description: NAPSI grades nails for both nail matrix psoriasis and nail bed psoriasis. The most affected fingernail was determined at Baseline and used for the analysis.
  Nail matrix psoriasis consists of any of the following: pitting, leukonychia, red spots in the lunula, or nail plate crumbling. Nail bed psoriasis is the presence or absence of onycholysis, splinter hemorrhages, oil drop (salman patch) discoloration or nail bed hyperkeratosis. Scoring for each is based on the following scale:
  * 0 = none;
  * 1 = present in 1/4 nail quadrants;
  * 2 = present in 2/4 nail quadrants;
  * 3 = present in 3/4 nail quadrants;
  * 4 = present in 4/4 nail quadrants.
  The sum of these two scores is the total score for the nail, and ranges from 0 (no nail psoriasis) to 8 (psoriasis in 4/4 nail quadrants). Change from Baseline is presented as a percentage of the Baseline value, calculated as: Week 24 value - Baseline value / Baseline value * 100. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population who had a NAPSI score ≥ 0 at the Baseline visit; last observation carried forward (LOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 22
percent change | -68.06 (34.134)

15. Other Pre Specified Outcome: Change From Baseline in Blood Cell Counts
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: × 10^9 cells/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
× 10^9 cells/L
  Platelets | -9.8 (55.51)
  White blood cells | 0.00 (2.248)
  Neutrophils | -0.446 (2.1341)
  Lymphocytes | 0.468 (0.6196)
  Monocytes | 0.006 (0.1992)
  Eosinophils | -0.036 (0.2905)
  Basophils | 0.013 (0.0602)

16. Other Pre Specified Outcome: Change From Baseline in Erythrocyte Sedimentation Rate
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Adalimumab
Number analyzed (Participants) | 46
mm/hour | -4.087 (9.8744)

17. Other Pre Specified Outcome: Change From Baseline in Alanine Aminotransferase
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
U/L | 2.8 (28.95)

18. Other Pre Specified Outcome: Change From Baseline in Aspartate Aminotransferase
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
U/L | 1.5 (16.81)

19. Other Pre Specified Outcome: Change From Baseline in Alkaline Phosphatase
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
U/L | -4.7 (14.84)

20. Other Pre Specified Outcome: Change From Baseline in Total Bilirubin
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
µmol/L | 0.5 (4.83)

21. Other Pre Specified Outcome: Change From Baseline in Creatinine
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
µmol/L | 2.1 (9.40)

22. Other Pre Specified Outcome: Change From Baseline in Blood Urea Nitrogen (BUN)
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
mmol/L | 0.42 (1.521)

23. Other Pre Specified Outcome: Change From Baseline in Uric Acid
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
µmol/L | -1.8 (66.52)

24. Other Pre Specified Outcome: Change From Baseline in Inorganic Phosphate
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
mmol/L | 0.061 (0.1900)

25. Other Pre Specified Outcome: Change From Baseline in Calcium, Sodium and Potassium
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
mmol/L
  Calcium | 0.005 (0.1035)
  Sodium | -0.8 (2.30)
  Potassium | 0.00 (0.435)

26. Other Pre Specified Outcome: Change From Baseline in Glucose
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
mmol/L | 0.12 (0.887)

27. Other Pre Specified Outcome: Change From Baseline in Albumin
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
g/L | 0.1 (2.87)

28. Other Pre Specified Outcome: Change From Baseline in Total Protein
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
g/L | -0.4 (3.91)

29. Other Pre Specified Outcome: Change From Baseline in Cholesterol
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
mmol/L | 0.045 (0.7723)

30. Other Pre Specified Outcome: Change From Baseline in Triglycerides
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
mmol/L | 0.194 (1.0007)

31. Other Pre Specified Outcome: Change From Baseline in High Sensitivity C-reactive Protein (hsCRP)
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
mg/L | -2.443 (5.2543)

32. Other Pre Specified Outcome: Change From Baseline in Urine pH
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pH units
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
pH units | 0.14 (0.663)

33. Other Pre Specified Outcome: Change From Baseline in Urine Specific Gravity
Description: Safety variables included laboratory data, vital signs and adverse events. Specific gravity is a measure of the amount of material dissolved in the urine. Specific gravity is the ratio of the density (mass of a unit volume) of a substance to the density (mass of the same unit volume) of a reference substance.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
ratio | 0.0003 (0.00792)

34. Other Pre Specified Outcome: Change From Baseline in Blood Pressure
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
mm Hg
  Systolic blood pressure | 0.9 (8.13)
  Diastolic blood pressure | -0.4 (7.03)

35. Other Pre Specified Outcome: Change From Baseline in Pulse
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
beats per minute | 0.2 (4.05)

36. Other Pre Specified Outcome: Change From Baseline in Respiratory Rate
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: respirations per minute
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
respirations per minute | -0.0 (1.33)

37. Other Pre Specified Outcome: Change From Baseline in Weight
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
kg | -0.18 (2.883)

38. Other Pre Specified Outcome: Change From Baseline in Body Temperature
Description: Safety variables included laboratory data, vital signs and adverse events.
Time Frame: Baseline and Week 24 (or Early Termination Visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees celsius
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
degrees celsius | -0.03 (0.191)

39. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence, which does not necessarily have a causal relationship with treatment.
  The investigator rated the severity of each AE as either:
  Mild: The AE is transient and easily tolerated; Moderate: The AE causes the participant discomfort and interrupts usual activities.
  Severe: The AE causes considerable interference with usual activities and may be incapacitating or life-threatening.
  A serious adverse event (SAE) is an AE that results in death, is life-threatening, results in or prolongs hospitalization, results in congenital anomaly, persistent or significant disability/incapacity, spontaneous or elective abortion, or requires intervention to prevent a serious outcome.
  Drug-related AEs are those assessed by the investigator as either probably or possibly related.
  Other malignancy excludes lymphoma, hepatosplenic T-cell lymphoma (HSTCL), leukemia, non-melanoma skin cancer (NMSC), and melanoma.
Time Frame: From the first dose of study drug until 70 days after the last dose (up to 33 weeks).
Measure: Number; unit: participants
Groups:
- Adalimumab: Number of participants with adverse events
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
participants
  Any adverse event | 14
  Serious adverse event | 0
  AE leading to discontinuation of study drug | 0
  Severe adverse event | 0
  Drug-related adverse event | 9
  Adverse event leading to death | 0
  Any infection | 7
  Any serious infection | 0
  Any opportunistic infection | 0
  Latent tuberculosis | 4
  Any lymphoma | 0
  Any non-melanoma skin cancer | 0
  Any other malignancy | 0
  Any demyelinating disorder | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 70 days after the last dose (up to 33 weeks).
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 14/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=50)
ANAEMIA (Blood and lymphatic system disorders) | 1
FURUNCLE (Infections and infestations) | 1
HERPES SIMPLEX (Infections and infestations) | 1
LATENT TUBERCULOSIS (Infections and infestations) | 4
ORAL HERPES (Infections and infestations) | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
RHINITIS (Infections and infestations) | 3
CONTUSION (Injury, poisoning and procedural complications) | 1
EXCORIATION (Injury, poisoning and procedural complications) | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1
BLOOD GLUCAGON INCREASED (Investigations) | 1
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1
RENAL COLIC (Renal and urinary disorders) | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.